CLINICAL TRIAL: NCT04943692
Title: Efficacy and Safety of Metformin Glycinate Compared to Metformin Hydrochloride on the Progression of Type 2 Diabetes
Acronym: COMETII
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Administrative decision of the investigation direction
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-30000-III-19(1)
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Metformin glycinate; Metformin hydrochloride; fasting glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — methionylglycine; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Metformin glycinate 1050 mg (Experimental): Metformin glycinate 1050 mg Orally twice a day.
  Interventions: Drug: Metformin glycinate
- Group B: Metformin hydrochloride 850 mg (Active Comparator): Metformin hydrochloride 850mg Orally twice a day.
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin glycinate — 1050 mg, tablets Administered orally, twice a day, for 12 months.
  Other Names: MET GLY
  Arms: Group A: Metformin glycinate 1050 mg
Drug: Metformin Hydrochloride — 850 mg, tablets. Administered orally, twice a day, for 12 months.
  Other Names: MET HYD
  Arms: Group B: Metformin hydrochloride 850 mg

SUMMARY:
Phase III study to evaluate the efficacy and safety of the treatment. Two-arm, prospective, longitudinal, double-blind, multicenter randomized clinical trial.

DETAILED DESCRIPTION:
Study to evaluate the efficacy and safety of treatment at 6 and 12 months with metformin glycinate at a dose of 2100 mg / day compared to metformin hydrochloride at a dose of 1700 mg / day on the progression of type 2 diabetes. To assess the change in HbA1c from baseline to 6 and 12 months of treatment (primary endpoint) in both groups. As secondary objectives, changes in fasting glucose levels from baseline, changes in results of the oral glucose tolerance test 2h from baseline, changes in HOMA-IR from baseline, changes in insulin levels, leptin, adipokines and proinflammatory cytokines, MCP-1, nitric oxide and PCr from baseline, changes in BMI from baseline and changes in lipid profile from baseline will be evaluated. A blinded interim analysis will be performed at 6 months of patient follow-up and a final analysis. Demographic data will be analyzed with mean, standard deviation, minimum and maximum. Efficacy analyzes will be carried out in the treated population (all treated patients, ATP), made up of all randomized patients who received at least one dose of the study treatment and who have a baseline measurement and at least one subsequent measurement.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years old.
* Type 2 diabetes according to ADA diagnostic criteria.
* Naive to treatment or who have previously been under oral hypoglycemic treatment (whatever it may be), as long as it has been suspended for a period of ≥6 weeks prior to the start of the study. - HbA1c ≥7.5% and <10.0%.
* In the case of women of childbearing age and with an active sexual life, the use of birth control methods is required; any of the following are accepted: barrier (male or female condom), non-hormonal intrauterine device, or bilateral tubal obstruction.
* That you agree to participate in the study and give written informed consent.

Exclusion Criteria:

* Patients with known current abuse or dependence (last 2 months) to substances such as alcohol (weekly consumption> 21 units of alcohol in men or> 14 units of alcohol in women) or recreational drugs.
* Body Mass Index <20 kg / m2 and> 35 kg / m2.
* Glomerular filtration estimated with the MDRD (Modification of Diet in Renal Disease) procedure through serum creatinine <60 ml / min / 1.72 m2.
* History of chronic liver disease or ALT (alanine aminotransferase) and / or AST (aspartate aminotransferase) ≥ 2 times the upper limit of normal, or GGT (Gamma glutamyl transpeptidase) ≥3 times the upper limit of normal.
* Chronic lung disease, causing dyspnea equivalent to a functional class ≥3 (NYHA) or requiring oxygen supplementation.
* Use of drugs that interact with biguanides.
* Other chronic diseases that limit survival or are associated with chronic inflammation such as: cancer, leukemia, lymphoma, lupus erythematosus, asthma, rheumatoid arthritis, or HIV (human immunodeficiency virus) infection.
* Pregnancy or positive pregnancy test, as well as women who are breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline, 6 and 12 months
  Assess change in HbA1c

SECONDARY OUTCOMES:
Changes in fasting glucose | Baseline, 6 and 12 months
  Determine the change in fasting glucose levels
Change in the 2-hour oral glucose tolerance curve | Baseline, 6 and 12 months
  Determine the change from baseline in the results of the 2-hour oral glucose tolerance curve
Changes to HOMA-IR (Homeostatic model assessment and Insulin resistance | Baseline, 6 and 12 months
  Determine change in HOMA-IR
Changes in insulin levels | Baseline, 6 and 12 months
  Determine the changes in insulin levels
Changes in leptin levels | Baseline, 6 and 12 months
  Determine the changes in leptin levels
Changes in adipokine levels | Baseline, 6 and 12 months
  Determine the changes in adipokine levels
Changes in proinflammatory cytokine | Baseline, 6 and 12 months
  Determine the changes in proinflammatory cytokine
Changes in levels of MCP-1 (monocyte chemoattractant protein 1) | Baseline, 6 and 12 months
  Determine the changes in levels of MCP-
Changes in nitric oxide levels | Baseline, 6 and 12 months
  Determine changes in nitric oxide levels
Changes in C-reactive protein levels | Baseline, 6 and 12 months
  Determine changes in C-reactive protein levels
Changes in body mass index | Baseline, 6 and 12 months
  Determine changes in body mass index
Incidence of adverse events | Baseline, 6 and 12 months
  Determine the incidence of adverse events that occurred during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Fanghänel Salmón, M.D, Principal Investigator — Clinica integral del paciente diabético y obeso; Manuel González Ortiz, M.D, Principal Investigator — Instituto de terapéutica experimental y clínica (INTEC); Joel Rodríguez Saldaña, M.D, Principal Investigator — Resultados médicos, desarrollo e investigación SC. (REMEDI); María L Sánchez Aldana Robles, M.D, Principal Investigator — Investigación Biomédica para el Desarrollo de Fármacos, S.A de C.V. (IBIOMED-GDL); Francisco G Padilla Padilla, M.D, Principal Investigator — Independent; Jorge V Yamamoto Cuevas, M.D, Principal Investigator — Clínica Villa Coapa La Vereda S.C.; Edmundo D Ríos Mejía, M.D, Principal Investigator — Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V. (IBIOMED-AGS); Luis M Román Pintos, M.D, Principal Investigator — Hospital Hispanos S.A. de C.V.; Víctor Bohórquez López, M.D, Principal Investigator — Oaxaca Site Management Organization SC. (Red OSMO); Santiago P Ramírez Díaz, M..D, Principal Investigator — Centro de Investigación Médica Aguascalientes (Red OSMO); José De la Cruz Tun Pech, M.D, Principal Investigator — Mérida Investigación Clínica (Red OSMO); Fernando J Lavalle González, M.D, Principal Investigator — Servicio de endocrinología Hospital Univertsitario, UANL
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander GC, Sehgal NL, Moloney RM, Stafford RS. National trends in treatment of type 2 diabetes mellitus, 1994-2007. Arch Intern Med. 2008 Oct 27;168(19):2088-94. doi: 10.1001/archinte.168.19.2088. PMID 18955637
- [Background] U.K. prospective diabetes study. II. Reduction in HbA1c with basal insulin supplement, sulfonylurea, or biguanide therapy in maturity-onset diabetes. A multicenter study. Diabetes. 1985 Aug;34(8):793-8. PMID 2862087
- [Background] Kahn SE, Haffner SM, Heise MA, Herman WH, Holman RR, Jones NP, Kravitz BG, Lachin JM, O'Neill MC, Zinman B, Viberti G; ADOPT Study Group. Glycemic durability of rosiglitazone, metformin, or glyburide monotherapy. N Engl J Med. 2006 Dec 7;355(23):2427-43. doi: 10.1056/NEJMoa066224. Epub 2006 Dec 4. PMID 17145742
- [Background] Hermann LS, Schersten B, Melander A. Antihyperglycaemic efficacy, response prediction and dose-response relations of treatment with metformin and sulphonylurea, alone and in primary combination. Diabet Med. 1994 Dec;11(10):953-60. doi: 10.1111/j.1464-5491.1994.tb00253.x. PMID 7895460
- [Background] Phung OJ, Scholle JM, Talwar M, Coleman CI. Effect of noninsulin antidiabetic drugs added to metformin therapy on glycemic control, weight gain, and hypoglycemia in type 2 diabetes. JAMA. 2010 Apr 14;303(14):1410-8. doi: 10.1001/jama.2010.405. PMID 20388897
- [Background] Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):854-65. PMID 9742977
- [Background] Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1577-89. doi: 10.1056/NEJMoa0806470. Epub 2008 Sep 10. PMID 18784090
- [Background] Tzoulaki I, Molokhia M, Curcin V, Little MP, Millett CJ, Ng A, Hughes RI, Khunti K, Wilkins MR, Majeed A, Elliott P. Risk of cardiovascular disease and all cause mortality among patients with type 2 diabetes prescribed oral antidiabetes drugs: retrospective cohort study using UK general practice research database. BMJ. 2009 Dec 3;339:b4731. doi: 10.1136/bmj.b4731. PMID 19959591
- [Background] Selvin E, Bolen S, Yeh HC, Wiley C, Wilson LM, Marinopoulos SS, Feldman L, Vassy J, Wilson R, Bass EB, Brancati FL. Cardiovascular outcomes in trials of oral diabetes medications: a systematic review. Arch Intern Med. 2008 Oct 27;168(19):2070-80. doi: 10.1001/archinte.168.19.2070. PMID 18955635
- [Background] Johnson JA, Simpson SH, Toth EL, Majumdar SR. Reduced cardiovascular morbidity and mortality associated with metformin use in subjects with Type 2 diabetes. Diabet Med. 2005 Apr;22(4):497-502. doi: 10.1111/j.1464-5491.2005.01448.x. PMID 15787679
- [Background] Kooy A, de Jager J, Lehert P, Bets D, Wulffele MG, Donker AJ, Stehouwer CD. Long-term effects of metformin on metabolism and microvascular and macrovascular disease in patients with type 2 diabetes mellitus. Arch Intern Med. 2009 Mar 23;169(6):616-25. doi: 10.1001/archinternmed.2009.20. PMID 19307526
- [Background] Tucker GT, Casey C, Phillips PJ, Connor H, Ward JD, Woods HF. Metformin kinetics in healthy subjects and in patients with diabetes mellitus. Br J Clin Pharmacol. 1981 Aug;12(2):235-46. doi: 10.1111/j.1365-2125.1981.tb01206.x. PMID 7306436
- [Background] Wang DS, Jonker JW, Kato Y, Kusuhara H, Schinkel AH, Sugiyama Y. Involvement of organic cation transporter 1 in hepatic and intestinal distribution of metformin. J Pharmacol Exp Ther. 2002 Aug;302(2):510-5. doi: 10.1124/jpet.102.034140. PMID 12130709
- [Background] Wilcock C, Bailey CJ. Accumulation of metformin by tissues of the normal and diabetic mouse. Xenobiotica. 1994 Jan;24(1):49-57. doi: 10.3109/00498259409043220. PMID 8165821
- [Background] Scheen AJ. Clinical pharmacokinetics of metformin. Clin Pharmacokinet. 1996 May;30(5):359-71. doi: 10.2165/00003088-199630050-00003. PMID 8743335
- [Background] Dunn CJ, Peters DH. Metformin. A review of its pharmacological properties and therapeutic use in non-insulin-dependent diabetes mellitus. Drugs. 1995 May;49(5):721-49. doi: 10.2165/00003495-199549050-00007. PMID 7601013
- [Background] Vidon N, Chaussade S, Noel M, Franchisseur C, Huchet B, Bernier JJ. Metformin in the digestive tract. Diabetes Res Clin Pract. 1988 Feb 19;4(3):223-9. doi: 10.1016/s0168-8227(88)80022-6. PMID 3359923
- [Background] Marathe PH, Wen Y, Norton J, Greene DS, Barbhaiya RH, Wilding IR. Effect of altered gastric emptying and gastrointestinal motility on metformin absorption. Br J Clin Pharmacol. 2000 Oct;50(4):325-32. doi: 10.1046/j.1365-2125.2000.00264.x. PMID 11012555
- [Background] Pacanowski MA, Hopley CW, Aquilante CL. Interindividual variability in oral antidiabetic drug disposition and response: the role of drug transporter polymorphisms. Expert Opin Drug Metab Toxicol. 2008 May;4(5):529-44. doi: 10.1517/17425255.4.5.529. PMID 18484913
- [Background] Wiernsperger NF, Bailey CJ. The antihyperglycaemic effect of metformin: therapeutic and cellular mechanisms. Drugs. 1999;58 Suppl 1:31-9; discussion 75-82. doi: 10.2165/00003495-199958001-00009. PMID 10576523
- [Background] Hoffmann J, Spengler M. Efficacy of 24-week monotherapy with acarbose, metformin, or placebo in dietary-treated NIDDM patients: the Essen-II Study. Am J Med. 1997 Dec;103(6):483-90. doi: 10.1016/s0002-9343(97)00252-0. PMID 9428831
- [Background] Schimmack G, Defronzo RA, Musi N. AMP-activated protein kinase: Role in metabolism and therapeutic implications. Diabetes Obes Metab. 2006 Nov;8(6):591-602. doi: 10.1111/j.1463-1326.2005.00561.x. PMID 17026483
- [Background] Standeven KF, Ariens RA, Whitaker P, Ashcroft AE, Weisel JW, Grant PJ. The effect of dimethylbiguanide on thrombin activity, FXIII activation, fibrin polymerization, and fibrin clot formation. Diabetes. 2002 Jan;51(1):189-97. doi: 10.2337/diabetes.51.1.189. PMID 11756340
- [Background] Gregorio F, Ambrosi F, Manfrini S, Velussi M, Carle F, Testa R, Merante D, Filipponi P. Poorly controlled elderly Type 2 diabetic patients: the effects of increasing sulphonylurea dosages or adding metformin. Diabet Med. 1999 Dec;16(12):1016-24. doi: 10.1046/j.1464-5491.1999.00201.x. PMID 10656230
- [Background] Pavlovic D, Kocic R, Kocic G, Jevtovic T, Radenkovic S, Mikic D, Stojanovic M, Djordjevic PB. Effect of four-week metformin treatment on plasma and erythrocyte antioxidative defense enzymes in newly diagnosed obese patients with type 2 diabetes. Diabetes Obes Metab. 2000 Aug;2(4):251-6. doi: 10.1046/j.1463-1326.2000.00089.x. PMID 11225659
- [Background] Beisswenger P, Ruggiero-Lopez D. Metformin inhibition of glycation processes. Diabetes Metab. 2003 Sep;29(4 Pt 2):6S95-103. doi: 10.1016/s1262-3636(03)72793-1. PMID 14502106
- [Background] Yamanouchi T, Sakai T, Igarashi K, Ichiyanagi K, Watanabe H, Kawasaki T. Comparison of metabolic effects of pioglitazone, metformin, and glimepiride over 1 year in Japanese patients with newly diagnosed Type 2 diabetes. Diabet Med. 2005 Aug;22(8):980-5. doi: 10.1111/j.1464-5491.2005.01656.x. PMID 16026361
- [Background] Brown JB, Conner C, Nichols GA. Secondary failure of metformin monotherapy in clinical practice. Diabetes Care. 2010 Mar;33(3):501-6. doi: 10.2337/dc09-1749. Epub 2009 Dec 29. PMID 20040656